CLINICAL TRIAL: NCT01600703
Title: Sitagliptin (®Januvia) Regulation of Intestinal and Hepatic Lipoprotein Particle and Hepatic Glucose Production in Humans
Brief Title: Sitagliptin Regulation of Intestinal and Hepatic Lipoprotein Particle and Hepatic Glucose Production in Humans
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Sitagliptin-REB-09-0428-B
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Hyperlipidemia
Keywords: Intestinal lipoprotein; Apolipoprotein B48 and apolipoprotein B100; Pancreatic clamp; DPPIV inhibitor
MeSH Terms: conditions — Hyperlipidemias | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): sitagliptin, 100mg, oral, single dose
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo, oral, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin, 100mg, oral, single dose
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — Placebo, oral, single dose
  Arms: Placebo

SUMMARY:
Recent studies in both animals and humans has demonstrated that the hormone GLP-1 (glucagon like peptide 1) reduces intestinal production of lipoprotein particles. The investigators therefore hypothesise that the drug sitagliptin which prevents the breakdown of GLP-1 will reduce intestinal lipoprotein production in humans. The investigators are unable to speculate whether sitagliptin will affect hepatic lipoprotein production because of lack of of data from animal studies or in vitro data. Sitagliptin is already an approved treatment for type 2 diabetes.

DETAILED DESCRIPTION:
Each subject will be studied twice 4-6 weeks apart in random order in this single blinded study. In study A they will receive a single dose of sitagliptin 100mg od. In study B they will receive placebo. A nasoduodenal tube will be sited under fluoroscopic guidance the day prior to the study. On the day of the study regular liquid formula (Great shake plus) will be infused from 4am through the tube to maintain a constant fed state. A pancreatic clamp (octreotide with replacement glucose, insulin and growth hormone) along with saline/sitagliptin will be started at 7am. From 9am an iv bolus of deuterated-glycerol (d5-glycerol) along with a regular infusion of deuterated leucine (L-[5,5,5-2H3]. Regular blood samples will be drawn to assess lipoprotein kinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 60 years
2. Body mass index 20 kg/m2 to 27 kg/m2
3. Hemoglobin above 130g/L.
4. Normal glucose tolerance in response to a 75g, 2-hr OGTT

Exclusion Criteria:

1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180) or proliferative retinopathy
3. History of diabetes or OGTT indicative of diabetes or impaired glucose tolerance.
4. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.
5. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH > 6 mU/l
6. Current addiction to alcohol or substances of abuse as determined by the investigator.
7. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
8. Taking any prescription or non-prescription medications at the time of the study
9. Having donated blood three months prior to and three months post study procedures
10. A pregnancy test will be performed 1 to 3 days prior to each study in all female subjects. Those who test positive for pregnancy will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Lewis, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Xiao C, Dash S, Morgantini C, Patterson BW, Lewis GF. Sitagliptin, a DPP-4 inhibitor, acutely inhibits intestinal lipoprotein particle secretion in healthy humans. Diabetes. 2014 Jul;63(7):2394-401. doi: 10.2337/db13-1654. Epub 2014 Feb 28. PMID 24584549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Local newspaper advertisement
Pre-assignment Details: 21 participants were enrolled in the study, however only 15 were started.
Groups:
- Placebo First, Then Sitagliptin; Sitagliptin First, Then Placebo: placebo, oral, single dose sitagliptin, 100 mg, oral, single dose
Period: First Intervention
Arm/Group | Placebo First, Then Sitagliptin | Sitagliptin First, Then Placebo
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Sitagliptin | Sitagliptin First, Then Placebo
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: placebo, oral, single dose sitagliptin, 100 mg, oral, single dose
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  Canada | 15
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (0.6)
Glucose Levels [Mean (Standard Deviation); unit: mmol/l] | 4.9 (0.1)
Triglyceride Levels [Mean (Standard Deviation); unit: mmol/l] | 1.2 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Apolipoprotein B48 Production Rate After Acute Oral Administration of 100mg Sitagliptin (Compared to Placebo)
Description: Apolipoprotein B48 turnover was measured in a 10-hour kinetic study with in vivo tracer techniques and mathematical modeling to calculate production rates. Studies were performed under conditions of a pancreatic clamp and a steady state fed state in volunteers receiving single oral dose of either 100mg sitagliptin or matching placebo.
Time Frame: 10 hours
Measure: Mean (Standard Error); unit: ug/kg/day
Groups:
- Sitagliptin: sitagliptin, 100 mg, oral, single dose
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 15 | 15
ug/kg/day | 122.9 (30.4) | 60.6 (12.2)

2. Secondary Outcome: Apolipoprotein B100 Production Rate After Acute Oral Administration of 100mg Sitagliptin (Compared to Placebo)
Description: Apolipoprotein B100 turnover was measured in a 10-hour kinetic study with in vivo tracer techniques and mathematical modeling to calculate production rates. Studies were performed under conditions of a pancreatic clamp and a steady state fed state in volunteers receiving single oral dose of either 100mg sitagliptin or matching placebo.
Time Frame: 10 hours
Measure: Mean (Standard Error); unit: mg/kg/day
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 15 | 15
mg/kg/day | 17.6 (1.8) | 20.4 (2.9)

ADVERSE EVENTS:
Time Frame: 10 hours
Arm/Group | Placebo | Sitagliptin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes